CLINICAL TRIAL: NCT02539095
Title: A Double-blind, Randomized, Post-marketing Surveillance to Evaluate the Efficacy of Intra-articular Collagen Injection in Patients With Knee Joint Pain Compared to Normal Saline Injection
Brief Title: Efficacy of Intra-articular Collagen Injection in Patients With Knee Joint Pain Compared to Normal Saline Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01CTZ
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Chondromalacia; Osteoarthritis; Traumatic Arthritis
Keywords: intra-articular injection; intra-articular collagen injection; collagen; knee joint pain
MeSH Terms: conditions — Cartilage Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cartizol, collagen injection (Experimental): Their eligibility to participate in the study is checked, and they are randomized either into the intra-articular collagen injection group based on a randomization table.
  Interventions: Device: CartiZol
- Normal Saline injection (Placebo Comparator): Their eligibility to participate in the study is checked, and they are randomized either into the (placebo) injection group based on a randomization table.
  Interventions: Device: Normal saline

INTERVENTIONS:
Device: CartiZol — The product, CartiZol, which contains absorbable collagen, is applied on the cartilage defect to stimulate the neovasculization and cell penetration and to assist the natural wound healing process. It supplements the defective or damaged cartilage. Place the needle on the tip of the syringe and inject the product into the articular cavity.
  Other Names: Intra articular collagen injection
  Arms: Cartizol, collagen injection
Device: Normal saline — 1. Supplementation of fluid and electrolytes (sodium or chlorine deficiency)
  2. Diluent for injection solution Place the needle on the tip of the syringe and inject the product into the articular cavity.
  Other Names: placebo
  Arms: Normal Saline injection

SUMMARY:
The primary objective of this study is to confirm the superiority of intra-articular collagen injection in patients with knee joint pain compared to the control group. 100mm VAS is used to measure the pain of the subjects 24 weeks after the procedure.

DETAILED DESCRIPTION:
This study is a double-blind clinical trial. Two hundred subjects has participated in it. The study is explained to the subjects, and they voluntarily choose to participate in it. Their eligibility to participate in the study is checked, and they are randomized either into the intra-articular collagen injection group or the normal saline (placebo) injection group based on a randomization table. They are asked to follow the guidelines of the investigators during the study and to visit the hospital five times, including for screening. At each visit, the subjects will undergo an examination with doctors, a medical examination by interview, and a blood test only when it is necessary to evaluate the safety and efficacy of the injection.

(*If the subjects performed the screening during the first visit on, the total number of his or her additional visits is four.)

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients aged 19 or older 2. Patients with knee joint pain due to chondromalacia, osteoarthritis (OA), or traumatic arthritis (TA) 3. Patients with 3 or lower score in the Kellgren-Lawrence grade 4. Patients with 40 mm or higher scores in the 100 mm VAS pain scale 5. Patients without significant pathological tests at their screening visit 6. Patients whose medication is confirmed within one week from their study enrolment and who agreed to maintain the medication dose during the study period if they need to keep taking it 7. When combination drugs are administered, considering the period of the drugs remaining in the body, patients who take the drugs stably for 2 weeks prior to participating in the trial (based on the screening, if it is confirmed that the patients took the drugs stably for 1 week prior to the screening, at the enrollment for injection, it should be assessed again, and the patients who are confirmed to have taken the drugs stably for 2 weeks prior to the trial could be registered).

  8. Patients who, after taking drugs for anesthetic purposes (provided to the subject after the injection) within one week after the intra-articular injection, agreed to take anti-inflammatory agents for no more than 5 consecutive days and for no more than 10 days in a month, and could stop taking the drugs within 2 days after the next visit even if the pain in the observation site becomes severe and thus additional drugs are required.

  9. Patients who agreed to use only the non-drug treatments (i.e., physiotherapy, osteopathy, and chiropractic therapy) allowed by the study investigators (Acupuncture is not allowed.) 10. Patients who agreed to receive the injection only in one knee when they feel pain on both knees (The other knee can be treated with prescribed drugs, but articular injections are not allowed.) 11. Patients or their representative (for adults) who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

* 1. Patients or their family members with a history of or an ongoing autoimmune disease 2. Patients with a history of anaphylactic response 3. Patients with hypersensitivity to grafting materials 4. Patients with hypersensitivity to porcine protein 5. Patient with grade 4 in the Kellgren-Lawrence grade 6. Patients with severe effusion 7. Patients who were injured severely or received injection in their affected knee within six months, which would make evaluation of the knee difficult 8. Patients with inflammatory arthritis such as rheumatoid arthritis, rupus arthrosis, or psoriatic arthritis 9. Patients who have gout or calcium pyrophosphate (pseudogout) disease that started within six months from the screening visit 10. Patients with a history of radiation therapy or cancer treatment within two years 11. Patients with diabetes 12. Patients with an infection that required hospitalization for antibiotics or the administration of antiseptic agents 13. Patients who have been undergoing adrenocortical hormone therapy 14. Patients with liver, heart, or kidney disease 15. Patients who had been infected with a virus 16. Patients who have a serious health condition that may affect the study results 17. Patients who are pregnant, breastfeeding, or planning to become pregnant 18. Patients who are considered inappropriate for participation in this study due to their condition (e.g., a mental illness) based on the investigator's judgment 8-15: The investigator can decide whether or not the patient will be administered the injection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Score change of 100 mm VAS | 24 weeks after injection
  The difference of the score of the investigational group and the control group at baseline and 24 weeks after injection will be calculated and analyzed

SECONDARY OUTCOMES:
Score change of WOMAC (Western Ontario and McMaster Universities) | at the screening visit and then 4, 12, and 24 weeks after injection
  The difference of the value of the affected knee of the investigational group and the control group at baseline, 4 weeks, 12 weeks, and 24 weeks after injection will be calculated and analyzed
Score change of SF-36 (36-ltem Short-Form Health Survey) | at the screening visit and then 4, 12, and 24 weeks after injection
  The difference of the value of the affected knee of the investigational group and the control group at baseline, 4 weeks, 12 weeks, and 24 weeks after injection will be calculated and analyzed
Score change of Satisfaction evaluation by patients | at 4, 12, and 24 weeks after injection
  The improvement level of the investigational group and the control group will be evaluated by patients at the completion of clinical trial according to the 5 grade evaluation table. The difference of the improvement level (excellent+good+ moderate/total) of the two groups obtained at the completion of clinical trial will be compared and analyzed by z-test. In addition, the improvement level at each time point will be compared and analyzed.
Score change of Satisfaction evaluation by physician in charge | at 4, 12, and 24 weeks after injection
  The improvement level of the investigational group and the control group will be evaluated by clinicians at the completion of clinical trial according to the 5 grade evaluation table. The difference of the improvement level (excellent+good+ moderate/total) of the two groups obtained at the completion of clinical trial will be compared and analyzed by z-test. In addition, the improvement level at each time point will be compared and analyzed.
Score change of Physical examination | at the screening visit and then 4, 12, and 24 weeks after injection
  The difference of the score of the affected knee of the investigational group and the control group at the times prior to injection, 4 weeks, 12 weeks and 24 weeks after injection will be calculated and analyzed
Score change of 100 mm VAS | at the screening visit and then 4 and 12weeks after injection
  The difference of the score of the investigational group and the control group at before injection, 4 weeks and 12 weeks after injection will be calculated and analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Young Wan Moon, MD, Principal Investigator — Samsung Medical Cente; Yong In, MD, Principal Investigator — The Catholic University of Korea; Han Jun Lee, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Kwang Jun Oh, MD, Principal Investigator — Kunkuk University Medical Center; Hwa Sung Lee, MD, Principal Investigator — The Catholic University of Yeouido St. Mary's Hospital
Locations (5):
- South Korea (5):
  - Chung-Ang University Hospital, Seoul, Seoul
  - Kunkuk University Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Seoul
  - The Catholic University of Yeouido St. Mary's Hospital, Seoul, Seoul